CLINICAL TRIAL: NCT06540183
Title: Percutaneous Intramyocardial Septal Radiofrequency Ablation for Drug-refractory Obstructive Hypertrophic Cardiomyopathy in Children and Adolescents: An Early Feasibility Study
Brief Title: Percutaneous Intramyocardial Septal Radiofrequency Ablation for Obstructive Hypertrophic Cardiomyopathy in Children
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20232356
Record Dates: First submitted 2024-07-22; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-10

CONDITIONS: Hypertrophic Cardiomyopathy, Obstructive
Keywords: Percutaneous Intramyocardial Septal Radiofrequency Ablation; children; hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous intramyocardial septal radiofrequency ablation — Percutaneous intramyocardial septal radiofrequency ablation (PIMSRA) is an innovative minimally invasive ablation treatment. Under the real-time transthoracic echocardiography guidance, a radiofrequency electrode needle is introduced into the hypertrophied interventricular septum via the percutaneous intramyocardial approach. Then the needle tip is pushed to the target region of the interventricular septal (IVS) basal segment 8 to 10 mm from the subaortic valve. The main objective of PIMSRA is to reduce ventricular septal hypertrophy and left ventricular outflow tract obstruction by means of thermal ablation.

SUMMARY:
The primary purpose of this study was to demonstrate the safety and efficacy of percutaneous intramyocardial septal radiofrequency ablation (PIMSRA) in children and assessed its performance and functional outcomes in the follow-up. This is an observational, single-arm, single-center study.

DETAILED DESCRIPTION:
The prevalence of hypertrophic cardiomyopathy (HCM) ranks second among cardiomyopathies in children. The prognosis of HCM has been previously demonstrated to be closely correlated with age. HCM in childhood is frequently associated with severe symptoms and high mortality rates, exhibiting a 36% higher incidence of malignant ventricular arrhythmias compared to adults, and being twice as likely to necessitate advanced heart failure therapies such as heart transplantation or left heart assist devices. Surgical septal myectomy can effectively help patients with drug-refractory symptoms but carries risks inherent to invasive procedures and requires expertise that is not universally available. Alcohol septal ablation is not recommended for applications in the young patient group.

Percutaneous intramyocardial septal radiofrequency ablation (PIMSRA) is a new method for the treatment of HCM using a special diagnosis and treatment device on the target area of the heart under the guidance of echocardiography. The method breaks through the worldwide problem of minimally invasive treatment of the myocardium on the beating heart, thus avoiding X-ray radiation and contrast agent damage. Previous research has illustrated the effectiveness and safety of PIMSRA for adult patients with obstructive HCM. We have found that PIMSRA results in sustained improvement in exercise capacity, persistent reduction in left ventricle outflow tract (LVOT) gradient, and sustained improvement in cardiac function.

This is an early feasibility study to evaluate the clinical safety and efficacy of PIMSRA in pediatric patients, as well as to assess postoperative cardiac function and exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertrophic obstructive cardiomyopathy
* Age younger than 18 years
* Resting or provoking left ventricular outflow tract gradient ≥ 50 mmHg
* Drug-refractory symptoms or intolerable to pharmaceutical therapies
* Heart function of New York Heart Association ≥ class II

Exclusion Criteria:

* Secondary left ventricular hypertrophy (LVH) related to subaortic stenosis or aortic stenosis
* Presence of concomitant heart disease requiring surgery
* Left ventricular ejection fraction <40%
* Cardiac resynchronization therapy within 3 months

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with obstructive HCM who remain severely symptomatic despite medical therapy or have LVOT obstruction (peak gradient ≥ 50mmHg) underwent percutaneous intramyocardial septal radiofrequency ablation from September 2020 to December 2023. A total of 16 consecutive children younger than 18 were included.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Safety composite outcome | 30 days
  The number of people who reach the composite safety outcome (the occurrence of at least one) of the following measured variables: 1) all-cause death; 2) heart failure; 3) ventricular fibrillation.
Feasibility outcome | 6 months
  The proportion of people with a peak left ventricle outflow tract gradient lower than 30 mmHg or decreased by more than 50%.

SECONDARY OUTCOMES:
Major surgery-related adverse events | 30 days
  Emergency surgery, severe pericardial tamponade, conduction block due to deviation in ablation range, surgery related ventricular septal perforation, stroke and malignant arrhythmias.
LVOT gradient | through study completion, an average of 2 years
  Left ventricular outflow tract gradient as measured by echocardiography.
Maximum interventricular septal thickness | through study completion, an average of 2 years
  Maximum septal thickness as measured by echocardiography.
New York Heart Association functional scale | through study completion, an average of 2 years
  New York Heart Association class, including grade I, grade II, grade III, grade IV. A higher grade means worse heart function.

CONTACTS AND LOCATIONS:
Overall Officials: Liwen Liu, Ph.D, M.D., Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu L, Li J, Zuo L, Zhang J, Zhou M, Xu B, Hahn RT, Leon MB, Hsi DH, Ge J, Zhou X, Zhang J, Ge S, Xiong L. Percutaneous Intramyocardial Septal Radiofrequency Ablation for Hypertrophic Obstructive Cardiomyopathy. J Am Coll Cardiol. 2018 Oct 16;72(16):1898-1909. doi: 10.1016/j.jacc.2018.07.080. PMID 30309466
- [Background] Zhou M, Ta S, Hahn RT, Hsi DH, Leon MB, Hu R, Zhang J, Zuo L, Li J, Wang J, Wang B, Zhu X, Liu J, Han Y, Li X, Xu B, Zhang L, Hou L, Han C, Liu J, Liu L. Percutaneous Intramyocardial Septal Radiofrequency Ablation in Patients With Drug-Refractory Hypertrophic Obstructive Cardiomyopathy. JAMA Cardiol. 2022 May 1;7(5):529-538. doi: 10.1001/jamacardio.2022.0259. PMID 35353129